CLINICAL TRIAL: NCT03555617
Title: A Phase 1, Open-Label, 2-Cohort Study to Assess the Single Dose Pharmacokinetics of Two Formulations of TD-1473 and to Assess the Effect of a High-Fat Meal and Itraconazole on the Pharmacokinetics of TD-1473 in Healthy Subjects
Brief Title: Food-effect, Drug-Drug Interaction (DDI), and Formulation Bridging Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 0174
Record Dates: First submitted 2018-06-01; First posted 2018-06-13 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Inflammatory Bowel Disease
Keywords: healthy volunteers; drug-drug interaction; itraconazole; CYP3A; P-gp; Inflammatory Bowel Disease; IBD; Irritable Bowel Syndrome; IBS
MeSH Terms: conditions — Inflammatory Bowel Diseases; Irritable Bowel Syndrome | interventions — izencitinib; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TD-1473 formulation bridging & food effect (Experimental): Subjects will receive, on Day 1 of each period, a single 100 mg oral dose of the tablet formulation of TD-1473 in the fed or fasted state, or the PIC formulation of TD-1473 in the fasted state, as part of a 3-period, crossover design.
  Interventions: Drug: TD-1473
- TD-1473 with Itraconazole (Experimental): Subjects will receive a single 100 mg oral dose of the tablet formulation of TD-1473 in the fasted state on Day 1 of Period 1. In Period 2, subjects will receive, in the fasted state, single oral doses of 200 mg itraconazole solution on Days -4 through 7 for a total of 11 days, with a single 100 mg oral dose of the tablet formulation of TD-1473 co-administered on Day 1.
  Interventions: Drug: TD-1473; Drug: Itraconazole
- TD-1473 without Itraconazole (Experimental): Subjects will receive a single 100 mg oral dose of the tablet formulation of TD-1473 in the fasted state on Day 1 of Period 1.
  Interventions: Drug: TD-1473

INTERVENTIONS:
Drug: TD-1473 — oral capsule/tablet, QD
Drug: Itraconazole — oral solution, QD
  Arms: TD-1473 with Itraconazole

SUMMARY:
This is a Phase 1, open-label, 2-cohort, food-effect, DDI, and formulation bridging study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 to 55 years old
* Male subjects must abstain from sexual intercourse or use a highly effective method of birth control
* Women of child bearing potential must have a negative pregnancy test and either abstain from sex or use a highly effective method of birth control
* Body Mass Index (BMI) 18 to 32 kg/m2
* Willing and able to give informed consent
* Additional inclusion criteria apply

Exclusion Criteria:

* Planning to conceive a child during the study or within 2 months after the last dose of study drug
* Is positive for hepatitis A, B or C, and/or HIV
* Has clinically significant abnormalities in baseline laboratory evaluations
* Subject has a clinically significant abnormal electrocardiogram (ECG)
* Participated in another clinical trial of an investigational drug (or medical device) within 30 days prior to screening or is currently participating in another trial of an investigational drug (or medical device)
* Additional exclusion criteria apply

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2018-07-15 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) in Plasma | Up to 8 days post-dose
Time to maximum observed concentration (tmax) in Plasma | Up to 8 days post-dose
Area under the concentration-time curve from hour 0 to the last measurable concentration (AUC0-last) in Plasma | Up to 8 days post-dose
Area under the concentration-time curve extrapolated to infinity (AUC0-inf) in Plasma | Up to 8 days post-dose
Apparent terminal elimination half-life (t1/2) in Plasma | Up to 8 days post-dose
Apparent clearance (Cl/F) in Plasma | Up to 8 days post-dose
Apparent volume of distribution (Vz/F) in Plasma | Up to 8 days post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No
Theravance Biopharma, Inc. will not be sharing individual de-identified participant data or other relevant study documents.